CLINICAL TRIAL: NCT04361851
Title: LCI-HEM-DRMM-DPEM-001: Phase II Study of Daratumumab-Pembrolizumab for Multiple Myeloma Patients With ≥ Three Prior Lines of Therapy
Brief Title: Study of Dara-Pembro for Multiple Myeloma Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment due to competing studies
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-HEM-DRMM-DPEM-001; 00043318 (Other: Advarra IRB)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Pembrolizumab and Daratumumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Experimental
  Other Names: KEYTRUDA

SUMMARY:
This is a phase II, single-arm, open-label study in subjects with relapsed and/or refractory multiple myeloma (RRMM) comparing Pembrolizumab (Pembro) in combination with Daratumumab (Dara) to the historical control of Daratumumab.

DETAILED DESCRIPTION:
Heavily pre-treated multiple myeloma patients who are treated with single agent daratumumab have been reported to have median PFS of 4 months. A median PFS of 4 months corresponds to an 8-month progression-free survival rate of 25% (based on the exponential survival distribution). For this population of patients treated with Daratumumab and Pembrolizumab, the aim is to improve the 8-month PFS rate to 50%. Thirty-three RRMM patients who have received ≥ 3 lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD) will be eligible for enrollment. Sixteen (16) subjects will be enrolled in the first stage, and if at least 5 of the 16 patients are alive and progression free at 8 months, an additional 17 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria Subjects must meet all of the following inclusion and exclusion criteria to participate in the trial.

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of ≤ 1.
4. Documented symptomatic/active multiple myeloma with measurable disease that has previously responded to therapy (partial response or better by IMWG criteria) and since relapsed or is refractory to the last line of therapy. Refractory disease is defined as evidence of progressive disease per IMWG criteria within 60 days (measured from the end of the last cycle) after completing treatment with the last anti-myeloma drug regimen.

   Note: measurable disease is defined as
   * Serum monoclonal protein level ≥ 0.5 g/dL for IgG, IgA, or IgM disease
   * Monoclonal protein or total serum IgD ≥ 0.5 g/dL for IgD disease
   * Urinary M-protein excretion of ≥ 200 mg over a 24-hour period
   * Involved free light chain level ≥ 10 mg/dL, along with an abnormal free light chain ratio
5. Subjects must have a documented history of relapsed and/or refractory multiple myeloma with 3 or more prior lines of therapy.
6. Subjects must have had prior exposure to daratumumab in one of the prior lines of therapy.
7. Prior cancer treatment, including chemotherapy and radiation therapy, must be completed at least 14 days prior to enrollment and the subject must have recovered from all reversible acute toxic effects of the regimen to their previous baseline or ≤ Grade 1. Exceptions include alopecia (all grades) and neuropathy (grade 1 with controlled pain, grade 2 without pain).
8. Demonstrate adequate organ function as defined below; all screening labs to be obtained within 3 days prior to initiating study treatment:

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
   * Platelets ≥ 75 x 109/L
   * Hemoglobin ≥ 8 g/dL or 4.96 mmol/L
   * Calculated creatinine clearance ≥ 30 mL/min/1.73m2
   * Corrected serum calcium ≤ 14.0 mg/dL
   * Serum total bilirubin ≤ 1.5 X ULN OR
   * Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study treatment. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

1. Subjects with active infection requiring systemic therapy such as known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) or HIV. (NOTE: at discretion of investigator, subjects with uncomplicated urinary tract infections may be eligible.)
2. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of trial participation, starting with consent through 120 days after the last dose of pembrolizumab and 3 months of last dose of daratumumab (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
3. Autologous stem cell transplantation within 12 weeks of cycle 1, day 1
4. History of previous or concurrent malignancy other than MM within the past 2 years. Exceptions include basal cell or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
5. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Known history of interstitial lung disease, known history of non-infectious pneumonitis that required steroids, current pneumonitis, known chronic obstructive pulmonary disease (COPD) with FEV1 ≤ 30% of predicted normal, known moderate or severe persistent asthma within the past 2 years, SpO2 ≤ 90%.
7. Has known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), with any neurologic symptoms resolved or stabilized without requirement of steroid treatment for at least 14 days prior to cycle 1, day 1.
8. Clinically significant cardiac disease including myocardial infarction within 6 months before cycle 1 day 1, or unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g. unstable angina, congestive heart failure NYHA class III-IV), clinically significant cardiac arrhythmia (NCI CTCAE grade ≥ 2).
9. Grade 2 peripheral neuropathy with associated pain or grade ≥3 peripheral neuropathy regardless of the presence of pain.
10. Plasma cell leukemia, Waldenstrom macroglobulinemia, POEMS syndrome, or amyloidosis.
11. Major surgery within 2 weeks before Cycle 1, Day 1. Subjects with prior surgery must be expected to have fully recovered from surgery during the time the subject is expected to receive treatment on study.
12. Prior exposure to an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 agent.
13. Severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
14. History of solid organ transplantation.
15. History of allogeneic stem cell transplantation.
16. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of cycle 1, day 1.
17. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1, Day 1.
18. Has a known history of active TB (Bacillus Tuberculosis).
19. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Cycle 1, Day 1.
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
8-Month Progression-Free Survival (PFS8) | 8 months
  PFS8 will be determined for each subject as a binary variable indicating whether or not the subject is alive and progression free at 8 months.

SECONDARY OUTCOMES:
Complete Response (CR) Rate | up to 5 years
  CR will be determined for each subject as a binary variable indicating whether or not the specific level of response was achieved.
Stringent Complete Response (sCR) Rate | up to 5 years
  sCR will be determined for each subject as a binary variable indicating whether or not the specific level of response was achieved.
Clinical Benefit Rate (CBR) | up to 5 years
  CBR (achieving a minimal response or better) will be determined for each subject as a binary variable indicating whether or not the specific level of response was achieved.
Overall Response Rate (ORR) | up to 5 years
  ORR (achieving a PR or better) will be determined for each subject as a binary variable indicating whether or not the specific level of response was achieved.
Time to First Response (TTFR) | up to 5 years
  TTFR is defined as the time from the start of study treatment to the time when the first occurrence of a MR or better was achieved.
Time to Best Response (TTBR) | up to 5 years
  TTBR is defined as the time from the start of study treatment to the time when the best response of MR or better was achieved.
Duration of Response (DOR) | up to 5 years
  DoR will be calculated for those subjects who achieve a PR or better and is defined as the time first occurrence of PR (or better) until the time of disease progression or death.
Progression-Free Survival (PFS) | up to 5 years
  PFS is defined as the duration of time from the initiation of study treatment to first occurrence of either progressive disease or death.
Overall Survival (OS) | up to 5 years
  OS is defined as the duration from initiation of study treatment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Usmani, MD, Principal Investigator — Wake Forest University Health Sciences